CLINICAL TRIAL: NCT03887195
Title: Evolution of Empathy and Emotional Intelligence During a Doctor-patient Relationship Training for 4th Year Medical Students
Brief Title: Evolution of Empathy and Emotional Intelligence During a Doctor-patient Relationship Training
Acronym: EMOREL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180446
Record Dates: First submitted 2019-03-15; First posted 2019-03-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Empathy; Emotional Intelligence
Keywords: empathy; emotional intelligence; Medical student; Educational program; Physician-Patient Relations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students: The clinical sample is made up of 501 students (male and female) in the 4th year of medicine at Paris Descartes University, participating at the obligatory training module during the 2018-2019 academic year : this constitutes the entire population concerned by the intervention.
  Interventions: Other: Training mandatory module about the therapeutic relationship

INTERVENTIONS:
Other: Training mandatory module about the therapeutic relationship — The training programme is composed by:
  * 2 lectures (optional)
  * 6 supervision sessions by Balint type groups (5 of which are mandatory);
  * 5 role-plays (all required);
  * 2 OSCE with patient actors (all required). This teaching is initiated by two lectures on the relationship, the awareness, the listening, the empathy, the therapeutic distance, and the personal impacts that affect the relationship.
  It included six sessions of Therapeutic Relation Training Groups inspired by the Balint groups. Five role-play sessions are also organized from January to May, the students could play the doctor or the patient. The scenarios are about the following themes: announcement of bad news; accompaniment of chronic disease; management of aggressiveness and hostility; etc. After the role-play, a feedback done by the teacher and the group helps to elaborate what has happened. Finally, a formative assessment will be made during the Clinical Objective Structured Examination.

SUMMARY:
Background: Empathic skills of medical students decrease during their studies. Besides, communication skills training is French context. In this context doctor-patient relationship training was built at Paris Descartes University for the 4th year medical students. Implementation of this training aims at maintaining or even increasing empathic and emotional skills of students.

Objective: to evaluate effectiveness of this training on medical students skills, knowledge and attitudes.

Methodology: Interventional and longitudinal monocentric study Pre/post-test auto-assessment for

* empathic skills score assessed with the Jefferson Scale of Physician Empathy- Medical Student Version (JSPE-MS)
* emotional intelligence's score assessed with the Emotional Expressivity Scale (EES)
* students' declarative knowledge of the doctor-patient relationship assessed with multiple choice question.

Post-test assessement for:

* empathic skills assessed by simulated patients with CARE grid during the Objective Structured Clinical Examination (OSCE).
* satisfaction auto-questionnaire.
* socio-demographic and education data.

DETAILED DESCRIPTION:
Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired.

Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures. (Limit: 32,000 characters)

Example:

Sudden out-of-hospital cardiac arrest (OOH-CA) remains a significant cause of death, in spite of recent declines in overall mortality from cardiovascular disease. Existing methods of emergency resuscitation are inadequate due to time delays inherent in the transport of a trained responder with defibrillation capabilities to the side of the OOH-CA victim. Existing Emergency Medical Services (EMS) systems typically combine paramedic Emergency Medical Technician (EMT) services with some level of community involvement, such as bystander cardiopulmonary resuscitation (CPR) training. Some communities include automated external defibrillators (AEDs) at isolated sites or in mobile police or fire vehicles. A comprehensive, integrated community approach to treatment with AEDs would have community units served by these volunteer non-medical responders who can quickly identify and treat a patient with OOH-CA. Such an approach is termed Public Access Defibrillation (PAD). Societal and medical developments have transformed the relationship between doctors and patients: several health system reforms, increasing time constraints that strongly impact the exchange between caregivers and patients, increasing of elderly population and rising prevalence of chronic diseases, complexification of therapeutic solutions, democratization of medical information through the media and internet; ... (1, 2).

Different studies point to the fact that there are some gaps in the field of communication.

The doctors themselves recognize that communication with their patients is one of the main difficulties in the practice of their profession, particularly for patients with chronic illness who do not adhere to care (9). The multiplication of blogs and discussion forums of young doctors on this topic is an example (10).

Some problems arising from this situation such as, inter alia, the non-compliance that is between 30% and 70%, according to different studies and the number of complaints which roses significantly (70-80% are estimated to be related to communications problems). In the mental health field, the style of communication influences the ability to detect a problem.

In view of these observations, medical and political authorities want to promote communication to enhance the doctor-patient relationship. The Royal College of Doctors and Surgeons of Canada have included it in one of the 7 Essential Skills that every doctor needs (with medical expertise, collaboration, management, health promotion, erudition and professionalism). In France, the law of 4 March 2002 on patients' rights and the quality of the healthcare system includes this point (33).

Numerous studies testify to the influence of communication in the area of health. A review of 21 studies, with a high methodological quality, shows that the quality of communication, during data collection and discussion of treatment, has a positive effect on patient health (35). The analyse shows that communication influences in decreasing order: emotional health, control of symptoms, physiological measures (such as blood glucose and blood pressure) and pain control (2).

Until recently, this learning was considered related to the practice (2). Different studies show the limits of practical experience (36-38). Other studies have shown the possibility of teaching communication skills to health professionals (37, 39-46).

In order to answer these questions, a training module on the therapeutic relationship was built at Paris Descartes University. This module is organized for 4th year medical students. The 4th year has been chosen because the students begin the externship, witch confronts students to the realities of their future profession: suffering, pain, death but also health inequalities, the precariousness and the power of the doctor. Paradoxically it is at this period that a fall of their empathy may be observed (48). The aim of this teaching is to develop the relational and communication skills (know-how and social skills). The pedagogical approach has been diversified to potentiate the contribution of this module on these three field: knowledge, well-being and know-how.

The training programme is composed by:

2 lectures (optional) 6 supervision sessions by Balint type groups (5 of which are mandatory); 5 role-plays (all required); 2 OSCE with patient actors (all required). This teaching is initiated by two lectures on the relationship, the awareness, the listening, the empathy, the therapeutic distance, and the personal impacts that affect the relationship. The courses are held in small groups to promote the personal investment of each student; they included six sessions of Therapeutic Relation Training Groups (each lasting one hour and a half) (49), from October 2018 to May 2019, inspired by the Balint groups (50). The effects of this groups are gradually clarified, especially in their psycho-affective aspects (projections, transference and countertransference, representations and beliefs, etc.).

Five role-play sessions are also organized from January to May, in one heure and half the students could play the doctor or the patient. The scenarios are about the following themes: announcement of bad news; accompaniment of chronic disease; management of a reluctant patient; management of so-called " abusive requests "; management of aggressiveness and hostility. After the role-play, a feedback done by the teacher and the group helps to identify and elaborate what has happened (about verbal and non-verbal communication), to point out the positive (and also negative ...) and suggest ways to improve.

Finally, a formative assessment will be made during the OCSE (Clinical Objective Structured Examination), two clinical stations are organized with simulated patients (professional actors). The feedback is then done by the patients themselves, supervised by the teacher who provided the role-play training.

Simulation allows the student to train in an environment close to reality, to understand the complexity and to reflect on his own thoughts, actions, emotions, as well as those of others. It allows working out a broad range of individual cognitive, relational, affective and psychomotor skills.

The Balint group is a space for discussion and reflection, supervised by an experienced professional. It is organized around clinical situations asking questions about the doctor-patient relationship. Many studies have investigated the impact of a typical Balint Group (GB), and more particularly, with general doctors, interns and medical students. GB reported a benefit for their professional life in terms of competence, strengthening their professional identity and sense of security (59) but not on job satisfaction (60).

The Balint Group increase psychological medicine skills and it also have a positive effect on the attitude towards patients with psychosomatic problems. The GB specifically augment significantly and uniquely the clinical empathy (66). It could be helpful to improve skills of medical students (71, 72) by promoting stress and anxiety management, self-awareness and a different view of the doctor-patient relationship (71).

Many studies show the impact of empathy on the doctor-patient relationship, a recent review (74) shows that empathy increases patient satisfaction. It improves the relationship skills by better control of patient anxiety, better communication (including psycho-social problems, better adherence to treatment and the reduction of certain symptoms). (74) For the doctor, improvement in empathy enhances the sense of personal accomplishment by improving his-own well-being (76).

However, during medical studies, clinical empathy decreases (48) especially from the third year, when students start to meet patients. A recent systematic review (77) explains this fall, which continues during the internship. This phenomenon also occurs in other health disciplines.

Neumann & al. hypothesize that the cause could be to live the experience of vulnerability at the beginning of the clinical practice; they also mention the role of idealized beliefs of the role of the doctor, as well as the high level of stress of some students (such as burnout, depression ...) (77).

The good influence of teaching on empathy has been shown, especially in hospital or in liberal cabinet (78, 79). However, insufficient lessons are organized to develop this skill.

A systematic review of 18 interventions to teach empathy to medical students, from 2003 to 2012, despite methodological biases, concludes that trainings to support student empathy are effective (80). A recent meta-analysis of 18 randomized controlled trials (81) confirms these findings.

Among the effective techniques, the simulation is highlighted as "experiential learning" and "theatre". Other studies also show the value of teaching empathy for interns (82) and doctors (83). Different pedagogies raise an interest in the teaching of empathy; including communication techniques (verbal and non-verbal), lessons based on the study of videotaped consultations, theoretical lessons in ethics and empathy, role playing and simulation with standardized patients (84), exchange groups and therapeutic relationship training groups (85), including Balint-type groups (86).

A first pilot study evaluating the evolution of the empathy of a part of the medical students, during the role plays was conducted during the 2017-2018 academic year, in order to evaluate the feasibility and relevance of this research, extended to the entire promotion of 4th year students.

The competency-based approach now constitutes a new frame of reference in education; who tries to go beyond pedagogy by objective (87). Emotional Intelligence is defined as "the ability to perceive, access and generate emotions to support thought, to understand emotions, and to promote emotional and intellectual growth."(88). As it now stands, the scientific literature has not been able to establish whether it was a personal trait, an acquired skill, or both (89). But a recent review indicates a correlation between medical education and the acquisition of emotional skills (69). It could be of great support in resolving some conflicting aspects of the doctor-patient relationship (69).

Indeed, the doctor-patient relationship is considered to be of significant "emotional risk"; because of the negative emotions expressed by the patient, such as pain, anxiety, despair ... (90). Paying attention to the emotions of the patient has a beneficial impact for both the patient and the doctor (prevention of the fall of empathy, greater professionalism, greater job satisfaction, and the last but not the least : well-being ...) (91, 92 ).

The increasing recognition of the notion of competence in the construction of medical professionalism (54), particularly in the area of doctor-patient relationship and communication (32), stimulate the organization of pedagogical devices. The FRT module attempts to respond to this approach. However, empathy and emotional intelligence appear as fundamental skills in the acquisition of these communicative and relational skills. This study aims to evaluate mainly the impact of this module of FRT on the maintenance or even the effective acquisition of certain skills and know-how (empathy and emotional intelligence) centrals in the construction of communication and relational skills.

In order to do that the analyse is focused to assess the evolution of the student's empathy score with the Jefferson Scale of Physician Empathy- Medical Student Version (JSPE-MS), and with the emotional intelligence's score by the Emotional Expressivity Scale (EES). Theses scores are collected at the beginning and the end of the module.

The empathic skills will be assessed by simulated patients with CARE grid during the Objective Structured Clinical Examination (OSCE).

This work investigates likewise the evolution of students' knowledge of the doctor-patient relationship with multiple choice questions.

At the end of the training students will be also asked to complete a satisfaction questionnaire. For the group baseline socio-demographic and education data will be collected.

This is a twofold study, quantitative and qualitative and the results about empathy and emotional intelligence are going to be put into perspective with the data about the acquisition of knowledge.

The statistical analysis evaluative intervention epidemiology:

-Quantitative : Scores collected before and after the training (JSPE-MS, EES,questionnaire about the knowledge) or just at the end of the module ( OSCE and satisfaction questionnaire)

The evolution of students' empathy will be evaluated by the JSPE-MS witch is a self-questionnaire assessing empathy specifically in the doctor-patient relationship. JSPE focuses more specifically on the cognitive component of empathy.

It is composed of 2O items, decomposable into 3 groups (Nuguyen Trong, 2016):

ten items focus on the " perspective talking " : adopting the patient's point of view (items 2, 4, 5, 9, 10, 13, 16, 17, 20) eight items relate to the "care component": the attention to the emotional experience of the patient (items 1, 7, 8, 11, 12, 14, 18, 19) two items represent "the ability to stand in the patient's shoes" (Items 3, 6) Each item is rated from 1 to 7 (Lickert scale). There is a specific version validated for students, the JSPE-MS that the investigators will use for this study.

The second self-related questionnaire is the EES (93), it is about the emotional expressivity. The French version was translated and submitted to the author. It evaluates the disposition to express emotions. This scale contains 17 proposals listing different forms of emotional expression, such as "I am able to cry in front of other people". The frequency of these situations, from "never true" to "always true" is rated from 1 to 6 on a Lickert scale.

Self-questionnaires about declarative knowledge are also submitted to students in order to complete the assessment of the skills acquired in this module, and to compare them with the empathic and emotional expressivity skills measured.

The multiple-response questionnaire it's proposed by the Sides platform, preparing students for the National Examination Grading (ECN) competition. The content will focus on part of the ECN Question No. 1, on "The doctor-patient relationship". Answers will be constructed from the National College of Psychiatry's reference system for psychiatry.

The last self-related questionnaire is submitted only at the end of the module, it's a student satisfaction questionnaire, taken from the WHO report on evaluation of educational devices (94). Student satisfaction is an important parameter in the acceptability of teaching and his investment (54). These results will be compared with the data of empathy and emotional expressiveness, to determine correlations.

At the end of the module, during the Objective Structured Clinical Examination (OSCE), students' empathy is measured by the evaluation by patients standardized. As the current pedagogical module can not allow pre / post-test evaluation of this measure, the post-test evaluation alone is proposed as representative of the skills of the cohort of students at the end of this module.

Finally, socio-demographic data will be collected, in order to relate the measures of empathy with these informations(96-98): age, sex, parents' level of education, living conditions of the students, internships done during the module, medical-psychiatric history (or has already done psychotherapy), specialty (s) desired after the internship: 1st, 2nd and 3rd choice.

The clinical sample is made up of 501 students (male and female) in the 4th year of medicine at Paris Descartes University, participating at the training module during the 2018-2019 academic year: this constitutes the entire population concerned by the intervention.

The study will be presented to students at the university's opening discours. The presentation will be made by one of the main pedagogical leaders of this module: Professor Jaury, who will show the benefits and "risks" of the study, the terms of participation (questionnaires) and the terms of consent or refusal An information note will be sent by email via the addresses transmitted to each student, with the same informations.

The questionnaires and a consent form will be made available to students on the Moodle platform, in the part where they access by their personal identifiers, before the beginning of the training and at the end of the module.

A new e-mail will be sent at the end of the year to the students to specify the modalities of this evaluation, its aim of research (and not sanctioning), to encourage to complete the self-questionnaires post-test, and to recall the benefits and risk of research, terms of consent and refusal.

The collection of pre-training data (JSPE-MS, EES) and socio-demographic data will be on the Moodle platform in the days preceding the start of the role plays.

The collection of post-training data will be done by filling the self-questionnaires immediately after the training OSCE, via the Moodle platform. A single entry will be made, via the Moodle platform, and will then be reported in a table for analysis, by Chiara Santini, one of the corresponding researchers.

Descriptive analyses will be performed to check for missing and / or outliers and to verify the normality of the variables and to decide which hypothesis tests to use.

All the data collected during the evaluation will be described in order to obtain a precise profile of the people participating in the study.

Quantitative variables will be described with confidence interval according to their mean, standard deviation, median, minimum and maximum.

The qualitative variables will be described according to their size and the percentage. The qualitative data analysis will follow a content analysis.

To check the differences between the two groups (pre and post-training), the analysis of variance, the Student's paired tests or the chi-squared test, will be done as some non-parametric tests (Kruskall-Wallis test or Wilcoxon-Mann-Whitney test ) may be used. Post hoc analysis will be conducted if necessary.

In order to know the relations between the quantitative variables the investigators will realize simple linear correlations (Pearson's R, or rho coefficient values for the Spearman correlation).

Multivariate analyses will be performed using multiple regressions. They will test the existence or not of a relationship between the predictive variables and the dependent variables considering the other confounding variables. The multivariate analyses will also make it possible to estimate whether each of the variables contributes significantly to the prediction of the dependent variable.

The statistics will be compiled and analyzed using the SPSS and R computer software. A significance level of 0.05 will be retained.

ELIGIBILITY:
Inclusion Criteria:

* Age > to 18 years old
* Undergraduate medical fourth-year student of Paris Descartes University
* Taking part in an obligatory doctor-patient relationship training
* French language
* Agreement

Exclusion Criteria:

Refusal of agreement

• Not speaking French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergraduate medical fourth-years student of Paris Descartes University
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Jefferson Scale of Physician Empathy- Medical Student Version (JSPE-MS) | The week before the beginning of intervention (first Balint group) and immediately after the end of the formative OSCE, up to 6 months later
  The evolution of students' empathy will be evaluated by the JSPE-MS which is a self-related questionnaire assessing empathy specifically in the doctor-patient relationship; JSPE focuses more specifically on the cognitive component of empathy.

SECONDARY OUTCOMES:
Emotional Expressivity Scale (EES) | The week before the beginning of intervention (first Balint group) and immediately after the end of the formative OSCE, up to 6 months later
  The emotional intelligence's score will be collected by the Emotional Expressivity Scale (EES). It evaluates the disposition to express emotions. This scale contains 17 proposals listing different forms of emotional expression. The frequency of these situations, from "never true" to "always true" is rated from 1 to 6 on a Lickert scale. The French version was translated and submitted to the author.
Multiple choice questions | The week before the beginning of intervention (first Balint group) and immediately after the end of the formative OSCE, up to 6 months later
  Students' declarative knowledge of the doctor-patient relationship will be assessed with multiple choice question
CARE grid | Immediately after the end of the formative OSCE, up to 6 months later
  Empathic skills will be assessed by simulated patients with CARE grid during the Objective Structured Clinical Examination (OSCE)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Aude PIOT, D, PhD candidate, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Céline Buffel du Vaure, MD, PhD, MCU, Study Chair — University of Paris 5 - Rene Descartes; Louis Baptiste Jaunay, MD, CCU, Study Chair — University of Paris 5 - Rene Descartes
Locations (1):
- Paris Descartes University, Sorbonne Paris City, Faculty of Medicine, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared with research team.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be completed at the end of data collection (at the end of june of 2019).
Access Criteria: All researchers involved in this research would be allowed to access to results.

REFERENCES:
- [Background] Richard C, Lussier M-T. La communication professionnelle en santé: Erpi; 2016.
- [Background] Starfield B, Wray C, Hess K, Gross R, Birk PS, D'Lugoff BC. The influence of patient-practitioner agreement on outcome of care. Am J Public Health. 1981 Feb;71(2):127-31. doi: 10.2105/ajph.71.2.127. PMID 7457681
- [Background] Maguire P, Fairbairn S, Fletcher C. Consultation skills of young doctors: I--Benefits of feedback training in interviewing as students persist. Br Med J (Clin Res Ed). 1986 Jun 14;292(6535):1573-6. doi: 10.1136/bmj.292.6535.1573. PMID 3719282
- [Background] Beckman HB, Markakis KM, Suchman AL, Frankel RM. The doctor-patient relationship and malpractice. Lessons from plaintiff depositions. Arch Intern Med. 1994 Jun 27;154(12):1365-70. PMID 8002688
- [Background] Marvel MK, Epstein RM, Flowers K, Beckman HB. Soliciting the patient's agenda: have we improved? JAMA. 1999 Jan 20;281(3):283-7. doi: 10.1001/jama.281.3.283. PMID 9918487
- [Background] Ormel J, Koeter MW, van den Brink W, van de Willige G. Recognition, management, and course of anxiety and depression in general practice. Arch Gen Psychiatry. 1991 Aug;48(8):700-6. doi: 10.1001/archpsyc.1991.01810320024004. PMID 1883252
- [Background] Arborelius E, Bremberg S. What does a human relationship with the doctor mean? Scand J Prim Health Care. 1992 Sep;10(3):163-9. doi: 10.3109/02813439209014056. PMID 1410945
- [Background] Beaulieu MD, Leclere H, Bordage G. Taxonomy of difficulties in general practice. Can Fam Physician. 1993 Jun;39:1369-75. PMID 8324406
- [Background] Novel A-S. Baptiste Beaulieu : " J'ai parfois l'impression que ma vie passe sans moi ". Le Monde.27.03.2015
- [Background] DiMatteo MR, Haskard-Zolnierek KB, Martin LR. Improving patient adherence: a three-factor model to guide practice. Health Psychology Review. 2012;6(1):74-91.
- [Background] DiMatteo MR. The physician-patient relationship: effects on the quality of health care. Clin Obstet Gynecol. 1994 Mar;37(1):149-61. doi: 10.1097/00003081-199403000-00019. No abstract available. PMID 8194205